CLINICAL TRIAL: NCT02112110
Title: Study of the Absolute Oral Bioavailability of BMS-791325 in Healthy Subjects
Brief Title: Absolute Bioavailability of BMS-791325
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: AI443-109; 2013-004645-17 (EudraCT Number)
Record Dates: First submitted 2014-04-08; First posted 2014-04-11 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-04

CONDITIONS: Hepatitis C Virus Infection
MeSH Terms: conditions — Hepatitis C | interventions — 8-cyclohexyl-N-((dimethylamino)sulfonyl)-1,1a,2,12b-tetrahydro-11-methoxy-1a-((3-methyl-3,8-diazabicyclo(3.2.1)oct-8-yl)carbonyl)cycloprop(d)indolo(2,1-a)(2)benzazepine-5-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMS-791325 (oral) and [13C]-BMS-791325 (IV) (Experimental): BMS-791325 single dose tablet orally and [13C]-BMS-791325 single dose solution intravenously on specific days
  Interventions: Drug: BMS-791325; Drug: [13C]-BMS-791325

INTERVENTIONS:
Drug: BMS-791325
Drug: [13C]-BMS-791325

SUMMARY:
The purpose of this study is to determine the absolute bioavailability of 150 mg oral dose of BMS-791325 relative to 100 µg IV infusion of [13C]-BMS-791325.

DETAILED DESCRIPTION:
Primary Purpose: Other: Protocol is designed to assess the absolute bioavailability of 150 mg (2x75 mg tablets) BMS-791325 administered orally

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

1. Healthy subjects as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations
2. Men and women ages 18 to 49 years, inclusive
3. Women of childbearing potential (WOCBP) must not be pregnant or breastfeeding

   * WOCBP and men who are sexually active with WOCBP must agree to follow protocol mandated instructions for method(s) of contraception during and after the study

Exclusion Criteria:

1. Any significant acute or chronic medical illness
2. Any current or recent gastrointestinal disease or surgery that could impact upon the absorption of study drug
3. Inability to tolerate oral medication
4. Inability to be venipunctured and/or tolerate venous access
5. Use of tobacco-containing or nicotine-containing products within 6 months
6. Recent (within 6 months of study drug administration) drug or alcohol abuse as defined in Diagnostic and Statistical Manual of Mental Disorders (4th Edition)(DSM IV), Diagnostic Criteria for Drug and Alcohol Abuse
7. Any of the following on 12-lead electrocardiogram (ECG) prior to study drug administration at screening or Day -1, confirmed by repeat

i)PR ≥ 210 msec

ii)QRS ≥ 120 msec

iii)QT ≥ 500 msec

iv)QTcF ≥ 450 msec

v)Second or third degree heart block

h) Positive urine screen for drugs of abuse

i) Positive blood screen for hepatitis C antibody, hepatitis B surface antigen, r HIV-1, -2 antibodies

j) Any of the following screening or Day -1 laboratory results outside the ranges specified below as defined by the laboratory, confirmed by repeat analysis:

i)Serum creatinine > upper limit of normal (ULN)

ii)Alanine aminotransferase (ALT) > ULN

iii)Aspartate aminotransferase(AST) > ULN

iv)Total bilirubin > ULN

k) History of any significant drug allergy (such as anaphylaxis or hepatotoxicity)

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Absolute oral bioavailability (F) of BMS-791325 | 48 hours from time of oral dosing
  Absolute bioavailability of 150 mg (2x75 mg tablets) BMS-791325 administered orally will be established by calculating the ratio of the dose normalized AUC(INF) of oral dose with that of 100 µg IV infused dose.

SECONDARY OUTCOMES:
Safety and tolerability of BMS-791325 by the occurrence of AEs and SAEs, abnormalities in vital sign measurements exceeding pre-defined thresholds, findings on ECGs and PEs, and abnormalities and marked abnormalities in clinical laboratory test. | Day 1 predose and 2 hours post-dose, Day 2 and Day 3
  Serious adverse events (SAEs)
  Adverse events (AEs)
  Physical examinations (PEs)
Maximum observed plasma concentration (Cmax) of BMS-791325 (oral dose) and [13C]-BMS-791325 (IV dose) | Pre-dose and at 0.5, 1, 1.5, 1.75, 1.97, 2, 2.125, 2.25, 2.5, 2.75, 3, 4, 5, 6, 8, 10, 12, 16, 24, 28, 32, 36 and 48 hours post oral dose
Time of maximum observed plasma concentration (Tmax) of BMS-791325 (oral dose) and [13C]-BMS-791325 (IV dose) | Pre-dose and at 0.5, 1, 1.5, 1.75, 1.97, 2, 2.125, 2.25, 2.5, 2.75, 3, 4, 5, 6, 8, 10, 12, 16, 24, 28, 32, 36 and 48 hours post oral dose
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC(0-T)) of BMS-791325 (oral dose) and [13C]-BMS-791325 (IV dose) | Pre-dose and at 0.5, 1, 1.5, 1.75, 1.97, 2, 2.125, 2.25, 2.5, 2.75, 3, 4, 5, 6, 8, 10, 12, 16, 24, 28, 32, 36 and 48 hours post oral dose
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC(INF)) of BMS-791325 (oral dose) and [13C]-BMS-791325 (IV dose) | Pre-dose and at 0.5, 1, 1.5, 1.75, 1.97, 2, 2.125, 2.25, 2.5, 2.75, 3, 4, 5, 6, 8, 10, 12, 16, 24, 28, 32, 36 and 48 hours post oral dose
Terminal plasma half-life (T-HALF) of BMS-791325 (oral dose) and [13C]-BMS-791325 (IV dose) | Pre-dose and at 0.5, 1, 1.5, 1.75, 1.97, 2, 2.125, 2.25, 2.5, 2.75, 3, 4, 5, 6, 8, 10, 12, 16, 24, 28, 32, 36 and 48 hours post oral dose
Total clearance (CLT) of [13C]-BMS-791325 (IV dose) | Pre-dose and at 0.5, 1, 1.5, 1.75, 1.97, 2, 2.125, 2.25, 2.5, 2.75, 3, 4, 5, 6, 8, 10, 12, 16, 24, 28, 32, 36 and 48 hours post oral dose
Volume of distribution at steady-state (Vss) of [13C]-BMS-791325 (IV dose) | Pre-dose and at 0.5, 1, 1.5, 1.75, 1.97, 2, 2.125, 2.25, 2.5, 2.75, 3, 4, 5, 6, 8, 10, 12, 16, 24, 28, 32, 36 and 48 hours post oral dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx